CLINICAL TRIAL: NCT07150572
Title: Evaluation of the Effect of Surgically Assisted Rapid Maxillary Expansion on Tooth Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 118115
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Maxillary Transverse Deficiency
Keywords: maxillary transverse deficiency; surgery asssisted rapid maxillary expansion; tooth color

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Under general anesthesia, the patients underwent a maxillary expansion procedure, during which the maxillary resistance sites were surgically released
  Interventions: Procedure: surgery assisted rapid maxillary expansion
- control group (No Intervention): no intervention

INTERVENTIONS:
Procedure: surgery assisted rapid maxillary expansion — Under general anesthesia, the patients underwent a maxillary expansion procedure, during which the maxillary resistance sites were surgically released
  Arms: Study Group

SUMMARY:
This prospective study aimed to evaluate effects of surgically assisted rapid maxillary expansion (SARME) on the color, maxillary anterior teeth by comparing them with untreated control group.

DETAILED DESCRIPTION:
In this study fifteen patients who underwent SARME and fifteen untreated control patients were included. Color measurements of the six maxillary anterior teeth were performed using a spectrophotometer. Periodontal health was assessed using the Gingival Index(GI), Probing Depth(PD), Plaque Index(PI), while pulp sensitivity was evaluated using an electric pulp tester(EPT). Color changes were calculated and fractal analysis was performed on CBCT images obtained evaluate the trabecular bone structure adjacent to the maxillary central incisors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the study group:

Young adult patients with completed growth and development,

Presence of maxillary transverse deficiency greater than 5 mm,

Patients with bilateral or unilateral posterior crossbite,

Absence of congenital tooth loss, fractures, restorative procedures, or root canal treatment in the maxillary arch,

Good patient cooperation.

Inclusion criteria for the control group:

Young adult patients with no history of orthodontic treatment,

Absence of congenital tooth loss, fractures, restorative procedures, or root canal treatment in the maxillary anterior teeth.

-

Exclusion Criteria:

* Exclusion criteria for both groups:

Patients consuming more than two cups of coffee or tea per day,

Patients who smoke,

Presence of systemic disorders that interfere with surgical procedures or bone metabolism,

Patients with craniofacial deformities or syndromic conditions,

Patients with poor cooperation.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Tooth color parameters | 17 months
  In this study patient who underwent SARME and untreated control groups teeth color were measured with spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Sunal Akturk, Assistant Professor, Study Chair — Saglik Bilimleri Universitesi; Gokmen Kurt, Professor, Study Chair — Bezmialem Vakif University; Fatma Derin Alpaydin, Research Assistant, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided